CLINICAL TRIAL: NCT01428414
Title: Multicenter, Randomized, Open-label Phase II Study to Compare the Efficacy and Safety of Trastuzumab and Paclitaxel Based Regimen Plus Carboplatin or Epirubicin as Neoadjuvant Therapy in HER2-positive Breast Cancer Patients
Brief Title: Efficacy and Safety Study of Trastuzumab and Paclitaxel Based Regimens to Treat HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhimin Shao (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Zhimin Shao, Professor and director of department of the Breast Cancer Institute, Fudan University, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML27770
Record Dates: First submitted 2011-08-28; First posted 2011-09-05 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: HER-2 Positive Breast Cancer
Keywords: HER2; Breast cancer; neoadjuvant chemotherapy; efficacy; safety
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel; Epirubicin; Injections; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trastuzumab+ Carboplatin+Paclitaxel (Active Comparator): Neoadjuvant treatment regimen:Trastuzumab,Carboplatin,Paclitaxel
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel; Drug: Carboplatin
- Trastuzumab+Epirubicin+Paclitaxel (Active Comparator): Neoadjuvant treatment regimen:Trastuzumab,Epirubicin,Paclitaxel
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel; Drug: Epirubicin

INTERVENTIONS:
Drug: Trastuzumab — 2 mg/kg, iv, d1,8,15(loading dose 4mg/kg wk1), qw
  Other Names: Herceptin
Drug: Paclitaxel — 75mg/m2, iv d1, 8,15. qw; 4-6 cycles
  Other Names: Taxol
Drug: Epirubicin — 75mg/m2, iv d1, q3w, 4-6 cycles
  Other Names: Epirubicin Hydrochloride for Injection
  Arms: Trastuzumab+Epirubicin+Paclitaxel
Drug: Carboplatin — AUC 2, qw, iv d1, 8,15. 4-6 cycles
  Other Names: CARBOPLATIN FOR INJECTION
  Arms: Trastuzumab+ Carboplatin+Paclitaxel

SUMMARY:
The purpose of the investigators study is to compare the efficacy and safety of combining trastuzumab and paclitaxel based regimen plus carboplatin or epirubicin as neoadjuvant therapy in Chinese HER2-positive breast cancer patients. 100 patients from multicenter would be randomly assigned into two treatment arms and receive neoadjuvant chemotherapy followed by operation and adjuvant treatment. The main end point of this study would be the efficacy and safety of the two treatment arms, and the trend of the two curves is anticipated.

DETAILED DESCRIPTION:
With the increased awareness and development of the diagnosis of breast cancer, more and more breast cancer is diagnosed at early. Amplification or overexpression, or both, of human epidermal growth factor receptor-2 (HER2, also known as ERBB2), a transmembrane receptor tyrosine kinase, is present in around 22% of early breast cancers, 35% of locally advanced and metastatic tumors, and 40% of inflammatory breast cancers, and is associated with aggressive disease and poor prognosis. The significant efficacy and good safety profile of Trastuzumab targeting HER 2 combination with chemotherapy as adjuvant treatment on EBC are accepted. Currently Trastuzumab has moved to Neoadjuvant treatment combined with chemotherapy based on many publications, among them pCR is accepted as primary endpoint to evaluate the efficacy of neoadjuvant therapy.

In the investigators study, Trastuzumab was concomitantly administered with different chemotherapies after randomization to determine the effect of this approach on the pathologic CR rates. 100 patients from multicenter would be randomly assigned into two treatment arms and receive neoadjuvant chemotherapy followed by operation and adjuvant treatment. Pathological complete response rate (pCR), disease free survival (DFS), response rates (RR), percentage of conserving breast surgery and adverse events including Serious AEs and non-serious AEs would be compared. The follow up time for each patients would be 3 years at most.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, presenting for the first time with invasive breast cancer, who have not received any previous treatment for an invasive malignancy
2. Aged ≥18 years and < 70 years with life expectancy > 12 months
3. Histologically confirmed invasive breast cancer (excluding inflammatory breast cancer) by core needle biopsy, staged II-III according to TNM Classification System, with no evidence of metastasis and tumor size ≥3 cm
4. HER2 positive confirmed by IHC 2+ and FISH positivity or IHC 3+
5. At least one measurable lesion according to RECIST criteria 1.1
6. Patients with a left ventricular ejection fraction(LVEF)≥55% by MUGA scan or echocardiography
7. ECOG PS 0-1
8. Willing to take biopsy before surgery and during chemotherapy and willing to take pre-operative chemotherapy and related treatment
9. Signed written informed consent; Able to comply with the protocol

Exclusion Criteria:

1. Patient is pregnant or lactating.
2. Women of child-bearing potential must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to take an adequate contraceptive measure
3. Previous treatment with chemotherapy or hormonal therapy or any prior therapy with an anti-HER2 therapy for any malignancy.
4. History of congestive heart failure, uncontrolled or symptomatic angina pectoris, arrhythmia or myocardial infarction
5. Other invasive malignancy (including second primary breast cancer) which could affect compliance with the protocol or interpretation of results. Patients who have been curatively treated and free of malignant disease for greater than 5 years are generally eligible
6. Inadequate bone marrow, hepatic and renal functions as evidenced by the following:

   * Neutrophil count of <1500/uL,
   * Platelet count of <100,000/uL.
   * Haemoglobin <10 g/dL.
   * Serum total bilirubin > 1.5*ULN (upper limit of normal),
   * ALT or AST > 2.5*ULN,
   * Alkaline phosphatase > 2.5*ULN,
   * Serum creatinine > 1.5*ULN.
7. Other serious illness or medical condition including:

   * Congestive heart failure (NYHA class II, III, IV) or history of documented congestive heart failure, unstable angina pectoris, myocardial infarction in the last 6 months, clinically significant valvular heart disease, or high-risk uncontrolled arrhythmias.
   * Patients with dyspnoea at rest due to malignant or other disease (e.g. pulmonary metastases with lymphangitis) or who require supportive oxygen therapy.
   * Active serious uncontrolled infections.
   * Poorly controlled diabetes mellitus.
8. Not willing to take pre-operative biopsy or neo-adjuvant therapy
9. Patients with psychiatric disorder or other disease leading to incompliance to the therapy
10. Known hypersensitivity to any ingredient of the regimen
11. Treatment with any investigational drug within 30 days before the beginning of treatment with study drug.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-08 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response rate | 3 years
  Percentage of complete pathological response, e.g. no microscopic evidence of residual invasive tumor cells in any resected specimens of the breast and/or axillary nodes.

SECONDARY OUTCOMES:
Disease free survival | 3 years at most
  Percentage of recurrence-free survival using Kaplan-Meier method, including subgroup analysis of DFS who complete 1-year trastuzumab treatment
Overall response rate | 3 years
  Percentage of clinical objective response using the RECIST scale
Percentage of conserving breast surgery | 3 years
  Percentage of conserving breast surgery
Safety | 3 years
  Incidence and severity of adverse events using the NCI-CTC scale 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ming Shao, MD, Principal Investigator — Fudan University
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Sikov WM, Dizon DS, Strenger R, Legare RD, Theall KP, Graves TA, Gass JS, Kennedy TA, Fenton MA. Frequent pathologic complete responses in aggressive stages II to III breast cancers with every-4-week carboplatin and weekly paclitaxel with or without trastuzumab: a Brown University Oncology Group Study. J Clin Oncol. 2009 Oct 1;27(28):4693-700. doi: 10.1200/JCO.2008.21.4163. Epub 2009 Aug 31. PMID 19720916
- [Background] Chang HR. Trastuzumab-based neoadjuvant therapy in patients with HER2-positive breast cancer. Cancer. 2010 Jun 15;116(12):2856-67. doi: 10.1002/cncr.25120. PMID 20564392
- [Background] Piccart-Gebhart MJ, Burzykowski T, Buyse M, Sledge G, Carmichael J, Luck HJ, Mackey JR, Nabholtz JM, Paridaens R, Biganzoli L, Jassem J, Bontenbal M, Bonneterre J, Chan S, Basaran GA, Therasse P. Taxanes alone or in combination with anthracyclines as first-line therapy of patients with metastatic breast cancer. J Clin Oncol. 2008 Apr 20;26(12):1980-6. doi: 10.1200/JCO.2007.10.8399. PMID 18421049
- [Background] Nistico C, Bria E, Cuppone F, Fornier M, Sperduti I, Carpino A, Pace A, Cognetti F, Terzoli E. Weekly epirubicin and paclitaxel with granulocyte colony-stimulating factor support in previously untreated metastatic breast cancer patients: a phase II study. Anticancer Drugs. 2007 Jul;18(6):687-92. doi: 10.1097/CAD.0b013e328035f863. PMID 17762397
- [Background] Gianni L, Eiermann W, Semiglazov V, Manikhas A, Lluch A, Tjulandin S, Zambetti M, Vazquez F, Byakhow M, Lichinitser M, Climent MA, Ciruelos E, Ojeda B, Mansutti M, Bozhok A, Baronio R, Feyereislova A, Barton C, Valagussa P, Baselga J. Neoadjuvant chemotherapy with trastuzumab followed by adjuvant trastuzumab versus neoadjuvant chemotherapy alone, in patients with HER2-positive locally advanced breast cancer (the NOAH trial): a randomised controlled superiority trial with a parallel HER2-negative cohort. Lancet. 2010 Jan 30;375(9712):377-84. doi: 10.1016/S0140-6736(09)61964-4. PMID 20113825
- [Background] Han S, Kim J, Lee J, Chang E, Gwak G, Cho H, Yang KH, Park S, Park K. Comparison of 6 cycles versus 4 cycles of neoadjuvant epirubicin plus docetaxel chemotherapy in stages II and III breast cancer. Eur J Surg Oncol. 2009 Jun;35(6):583-7. doi: 10.1016/j.ejso.2009.01.002. Epub 2009 Feb 5. PMID 19195817